CLINICAL TRIAL: NCT06540170
Title: Feasibility and Acceptability of a Personalized Self-care Support Program for Primary Care Patients With Diabetic Foot Ulcer
Brief Title: A Personalized Self-care Support Program for Primary Care Patients With Diabetic Foot Ulcer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Healthcare Group Polyclinics (Other Government)
Collaborators: Nanyang Technological University (Other)
Responsible Party: Principal Investigator, Julia Zhu Xiaoli, Senior Nurse Clinician Wound Management, National Healthcare Group Polyclinics
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022/00895
Record Dates: First submitted 2024-07-27; First posted 2024-08-06 (Actual); Results first posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Foot Ulcer
Keywords: Diabetic foot ulcer; self-care support; Motivational interviewing
MeSH Terms: conditions — Foot Ulcer; Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Single-group pre-intervention and post-intervention comparison
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Other): Eligible and willing participants will be invited to participate in the program and receive three 30-minute face-to-face sessions (once every 2 weeks) within 6 weeks of enrolment.
  Interventions: Behavioral: A personalised self-care support program

INTERVENTIONS:
Behavioral: A personalised self-care support program — A personalized care program consists of three 30-minute face-to-face sessions (once every 2 weeks) after patients' routine wound dressings to enhance self-efficacy, support emotional adjustments, and DFU self-care.

SUMMARY:
This clinical trial aims to learn if a personalized self-care program supporting self-care and Healing through Empowerment and Active Listening (HEALing), is acceptable to patients with diabetic foot ulcer (DFU) and wound care nurses, and is feasible to deliver supportive self-care for primary care patients living with DFU.

The main questions it aims to answer are:

* Is the personalized self-care improvement program acceptable to patients with diabetic foot ulcer (DFU) and wound care nurses to deliver?
* Is the personalized self-care improvement program feasible for supportive self-care for primary care patients living with DFU? Researchers will compare pre-intervention to post-intervention to see if the personalized self-care improvement program works to support self-care management for patients with DFU.

Participants will:

-receive three 30-minute face-to-face intervention sessions every 2 weeks within 6 weeks after their routine wound care dressing.

DETAILED DESCRIPTION:
This study aims to assess the potential benefit(s) of a personalized intervention integrating motivational interviewing (MI) with positive psychological skills for supportive self-care among patients with diabetic foot ulcers.

A single-arm pilot feasibility study using a mixed-method approach will be conducted between Aug 2024 and February 2025. 30 participants will be recruited from nurse-led wound clinics in a large primary care sector and selected according to the inclusion criteria. Participants will receive three 30-minute face-to-face sessions of an MI-based personalized care program over 6 weeks to support DFU self-care coping behaviors.

The primary outcomes include the feasibility of recruitment and the acceptability of the proposed personalized intervention. Feasibility will be assessed based on recruitment and 4 weeks retention of participants from last intervention session through examination of screening logs and follow-up completion. Acceptability to patients and healthcare professionals (HCPs) will be evaluated using semi-structured individual interviews.

The secondary outcomes include patient-reported outcome measures (PROM) consisting of DFU self-care behaviors, self-efficacy, psychological determinants, and clinical endpoints such as foot skin conditions and glycemic control (measured by HbA1C). The results will be evaluated by comparing baseline and post-intervention data collected at week 0 and week 4 from last intervention session, for any differences in PROMs and clinical outcomes. Differences in PROMs between the two time points will be assessed using univariable analyses such as the chi-square test for categorical variables and independent samples t-test or analysis of variance (ANOVA) for continuous variables where appropriate.

Semi-structured face-to-face individual qualitative interviews will be conducted at the end of the pilot trial to provide insight into peoples' experiences of participation in the intervention. Data will be analyzed thematically.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetes and DFU aged 21 years or above receiving treatment and wound care at National Healthcare Group Polyclinics
* HCPs, who are aged 21 years or above with a patient-facing role working in delivering program (only for qualitative interviews)

Exclusion Criteria:

* Patients have a diagnosis of critical lower limb ischemia, active osteomyelitis, Charcot foot, cognitive/psychiatric diagnoses, and hearing or vision impairment.
* Pregnant women will be excluded from the study for both patient and HCP groups

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2024-08-13 (Actual); Primary Completion 2025-01-11 (Actual); Study Completion 2025-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia Xiaoli Zhu, Principal Investigator — National Healthcare Group Polyclinics Singapore
Locations (1):
- National Healthcare Group Polyclinics, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhu X, Lee ES, Chan FHF, Yin R, Lim PXH, Koh RWS, Judith C, Wei L, Li S, Phrommarad P, Chin GHY, Lim VH, Low RSY, Chen YC, Griva K. Feasibility and acceptability of a personalised self-care support programme for primary care patients with diabetic foot ulcers delivered by wound care nurses: the HEALing study protocol. BMJ Open. 2025 Oct 7;15(10):e098024. doi: 10.1136/bmjopen-2024-098024. PMID 41062140

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm Study: Single-arm study: pre- and post-intervention
Period: Overall Study
Arm/Group | Single Arm Study
Started | 29
Completed | 26
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: Patients with diabetic foot ulcers receiving wound care at the participating clinics
Arm/Group | Single Arm Study
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 26
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Singapore | 26

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Recruiting and Retaining
Description: The number of patients recruited to the study and retained at the end of the study period will be documented.
Time Frame: 4 weeks post-intervention from baseline.
Population: 3 patients withdrew from the study due to changes to their healthcare institutions (e.g., from primary care settings to secondary/tertiary settings).
Measure: Count of Participants; unit: Participants
Groups:
- Single Arm: Eligible and willing participants will be invited to participate in the program and receive three 30-minute face-to-face sessions (once every 1-2 weeks) within 3-6 weeks of enrolment.
  A personalised self-care support program: A personalized care program consists of three 30-minute face-to-face sessions (once every 1-2 weeks) after patients' routine wound dressings to enhance self-efficacy, support emotional adjustments, and DFU self-care.
Arm/Group | Single Arm
Number analyzed (Participants) | 29
Participants | 26

2. Primary Outcome: Acceptability of the Intervention
Description: Participants will be interviewed to determine the acceptability of the intervention.
Time Frame: 4 weeks post-intervention from baseline.
Population: Participants with diabetic foot ulcers receiving wound care at the participating primary clinics
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Study
Number analyzed (Participants) | 29
Participants | 26

3. Secondary Outcome: Patients' Adherence to Foot Self-care Behaviour
Description: Measured using the 7-item Diabetes Foot Self-Care Behavior Scale. All items on the scale are rated on a 5-point Likert-type scale. The higher scores represent better foot self-care behaviors. The minimum value is 7 and the maximum is 35.
Time Frame: 4 weeks post-intervention from baseline.
Population: Participants with diabetic foot ulcers receiving wound care at the participating primary care clinics (excluding 3 withdrawals due to changes to primary care institutions)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm Study
Number analyzed (Participants) | 26
score on a scale | 20.2 (3.8)

4. Secondary Outcome: Patients' Foot Care Confidence (Self-efficacy)
Description: Measured using the 12-item Foot Care Confidence Scale. All items on the scale are rated on a 5-point Likert-type scale. The higher scores represent better foot care confidence. The minimum value is 12 and the maximum value is 60.
Time Frame: 4 weeks post-intervention from baseline.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm Study
Number analyzed (Participants) | 26
score on a scale | 32.7 (4.3)

5. Secondary Outcome: Patients' Illness Belief
Description: Measured using the 8-item Brief Illness Perception Questionnaire, each item is rated on a 0-10 scale, with higher scores indicating a more threatening perception of the illness.
  The total score is calculated by summing the scores of all eight items where items 3, 4, and 7 are inversed. The possible range of scores is 0 (minimum value)-80 (maximum value). Higher scores indicate worse illness perception.
Time Frame: 4 weeks post-intervention from baseline.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 26
score on a scale | 47.9 (10)

6. Secondary Outcome: Patients' Perceptions of Autonomy Support
Description: Measured using the 6-item Health Care Climate Questionnaire that patients rate items on a 7-point Likert scale (1 = not at all true, 7 = very true). The minimum value is 1 and the maximum value is 7. The higher score represents greater autonomy support.
Time Frame: 4 weeks post-intervention from baseline.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm Study
Number analyzed (Participants) | 26
score on a scale | 3.5 (0.9)

7. Secondary Outcome: Patients' Diabetes Distress
Description: Measured using Diabetes Distress Scale consists of 17 items with four subscales including emotional burden, physician-related distress, regimen-related distress, and interpersonal distress. All items were rated on a 6-point Likert scale. The minimum value is 1 and the maximum value is 6. The higher score indicates greater distress.
Time Frame: 4 weeks post-intervention from baseline.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm Study
Number analyzed (Participants) | 26
score on a scale | 3.5 (0.9)

8. Secondary Outcome: Patients' Knowledge of Recognizing Wound Deterioration
Description: Measured using Warning Signs of Diabetic Foot Ulcer Deterioration Questionnaire comprising of 12 items. Each item with the correct answer obtains a score of 1. The minimum score is 0 and the maximum value is 12. The higher scores represent better knowledge.
Time Frame: 4 weeks post-intervention from baseline.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm Study
Number analyzed (Participants) | 26
score on a scale | 7.7 (2.0)

9. Secondary Outcome: Patients' Quality of Life
Description: Measured using EQ-5D-5L that is self-reported by patients and consists of two parts: a descriptive system and a visual analogue scale. The visual analogue scale for imaginative health state is used for the pilot study. The minimum value is 0 and the maximum value is 100. The higher score represents the better 0 imaginative health state.
Time Frame: 4 weeks post-intervention from baseline.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Arm Study
Number analyzed (Participants) | 26
units on a scale | 57.3 (15.2)

10. Secondary Outcome: HbA1c
Description: HbA1c for participants who have completed the program.
Time Frame: 4 weeks post-intervention from baseline.
Population: Participants with an active DFU receiving wound care at the participating clinics
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | Single Arm Study
Number analyzed (Participants) | 19
mmol/mol | 83 (42)

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed (as this is a self-care education intervention with no risk of adverse event)
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed
Groups:
- Single Arm Study: All participants were assigned to a single intervention group receiving the programme in addition to standard diabetic foot ulcer care. No control or comparison group was included.
Arm/Group | Single Arm Study
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-10): https://cdn.clinicaltrials.gov/large-docs/70/NCT06540170/Prot_SAP_000.pdf